CLINICAL TRIAL: NCT06935032
Title: Evaluation of Mandibular Soft Tissue Changes in Patients Using Functional Appliances
Brief Title: Functional Appliance Effects on Mandibular Soft Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Seda Sağoğlu, Research Assistant / Principal Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/351
Record Dates: First submitted 2025-04-04; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Mandibular Retrognathism
Keywords: : Functional appliances; soft tissue change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Class II Division I malocclusion caused by mandibular retrognathia (Experimental): Class II Division I patients treated with the Twin Block appliance
  Interventions: Device: Twin block appliance
- Class II Division II malocclusion caused by mandibular retrognathia (Experimental): Class II Division II patients treated with the Twin Block appliance
  Interventions: Device: Twin block appliance
- Skeletal Class I patients (Experimental): Class I patients who received fixed treatment
  Interventions: Other: Fixed orthodontic treatment

INTERVENTIONS:
Device: Twin block appliance — An appliance that facilitates forward positioning of the mandible and soft tissues
  Arms: Class II Division I malocclusion caused by mandibular retrognathia; Class II Division II malocclusion caused by mandibular retrognathia
Other: Fixed orthodontic treatment — Patients undergoing orthodontic treatment with fixed appliances
  Arms: Skeletal Class I patients

SUMMARY:
This study aimed to evaluate the changes in mandibular and cervical soft tissues in Class II patients with mandibular retrognathia treated with the Twin Block appliance, compared to skeletal Class I patients without functional treatment, using profile photographs and cephalometric films. Sixteen patients with Class II Division 1, fifteen with Class II Division 2, and fifteen with skeletal Class I malocclusion were included. Measurements were performed at the beginning of treatment and after functional therapy. In the Class II Div 1 group, most parameters showed significant reductions, except for neck length and jaw tip contour. In the Class II Div 2 group, only the Sm-E plane measurement remained unchanged, while the control group showed minimal changes. Between-group comparisons indicated significant improvements in cervicomental angle, lip-jaw-throat angle, and other lower face soft tissue parameters, especially in Class II Division 1 patients. The findings suggest that Twin Block therapy effectively improves both skeletal and soft tissue profiles, with more pronounced soft tissue enhancement in Class II Division 1 cases.

DETAILED DESCRIPTION:
This retrospective study aims to investigate the changes in the mandibular and cervical soft tissues of patients with Class II malocclusion and mandibular retrognathia treated with the Twin Block appliance. The study includes patients treated in the Department of Orthodontics, Faculty of Dentistry, XXXX University, between 2021 and 2023. Ethical approval was obtained from the relevant ethics committee (Decision No: 2023/351), and informed consent was secured from all participants and their parents.

A total of 46 individuals were included: 16 patients with Class II Division I malocclusion, 15 with Class II Division II malocclusion, and 15 control subjects with skeletal Class I malocclusion. All patients in the treatment groups were in the growth spurt phase (CVMS3-S4) and received Twin Block therapy full-time for 12 months. The control group received fixed orthodontic treatment without functional appliances.

Profile photographs and lateral cephalometric radiographs were obtained at the beginning of treatment (T1) and after 1 year of therapy (T2), using a standardized protocol in natural head position (NHP). Measurements were performed digitally using Dolphin Imaging software. The study assessed angular parameters such as the submental-facial angle, cervicomental angle, lip-jaw-throat angle, and Sm-E plane angle from photographs, as well as linear measurements from cephalometric radiographs, including throat length, jaw tip contour, soft tissue pogonion thickness, soft tissue menton thickness, and lower lip-pogonion distance.

Sample size was determined via power analysis, which indicated that 15 patients per group were sufficient to detect clinically meaningful differences. To ensure measurement reliability, cephalometric analyses were repeated, and intra-observer reliability was confirmed with an intraclass correlation coefficient (ICC) of 0.924.

Statistical analyses were conducted using R software. Paired t-tests were employed for within-group comparisons, while independent t-tests and ANOVA with Tukey's post hoc tests were used for intergroup comparisons. Mixed-effects models and chi-square tests were utilized where appropriate. A significance level of p < 0.05 was adopted for all analyses.

This study was designed to contribute to the understanding of how Twin Block functional appliance therapy influences the morphology of the mandibular and cervical soft tissues, using both photographic and radiographic assessments in a growing patient population.

ELIGIBILITY:
Inclusion Criteria:

* having Class II malocclusion caused by mandibular retrognathia (ANB > 4°, SNB<78°),
* exhibiting horizontal and/or normal growth pattern (SN-GoGn=32 ±6),
* having profile photographs and cephalometric radiographs taken in the NHP (using the self-balance method one of the dynamic approaches for determining NHP)15,
* not requiring rapid maxillary expansion,
* not having increased initial lower incisor inclination on lateral cephalometric radiographs,
* Class II Division 2 patients presenting with ≥4 mm deepbite and the absence of any prior upper incisor protrusion methods,
* the control group individuals were required to have a skeletal Class I pattern (ANB angle between 0-4°) without any dental deficiencies.

Exclusion Criteria:

* previous orthodontic treatment,
* presence of craniofacial anomalies involving the jaw and/or teeth,
* severe facial asymmetry

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Patients treated with the Twin Block appliance | 12 month
  The changes in certain angular (degrees) and linear (millimeters) measurements may be considered favorable for the mandibular soft tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Sağoğlu, Principal Investigator — Konya Necmettin Erbaka University Faculty of Dentistry
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Malkoc S, Demir A, Uysal T, Canbuldu N. Angular photogrammetric analysis of the soft tissue facial profile of Turkish adults. Eur J Orthod. 2009 Apr;31(2):174-9. doi: 10.1093/ejo/cjn082. Epub 2008 Dec 8. PMID 19064675